CLINICAL TRIAL: NCT05348161
Title: Dynamic Multiomics Evaluation of Anti-HER2 and Immunotherapy in HER2 Positive Gastric Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, Professor, Peking University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CGOG-HER2-1001
Record Dates: First submitted 2022-01-29; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2021-12

CONDITIONS: HER2 Positive Advanced Gastric Cancer
MeSH Terms: interventions — Tissue Banks

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anti-HER2 & Immunotherapy (Other): Advancd gastric cancer patients received anti-HER2 & immunotherapy ± chemotherapy
  Interventions: Procedure: Samples including blood and tissue collection; Procedure: CTC detection; Procedure: ctDNA detection; Procedure: 10×genomics single cell RNA sequence; Procedure: Whole exon sequence; Procedure: Proteomics detection
- Anti-HER2 (Other): Advancd gastric cancer patients received anti-HER2 ± chemotherapy.
  Interventions: Procedure: Samples including blood and tissue collection; Procedure: CTC detection; Procedure: ctDNA detection; Procedure: 10×genomics single cell RNA sequence; Procedure: Whole exon sequence; Procedure: Proteomics detection

INTERVENTIONS:
Procedure: Samples including blood and tissue collection — Tissue and peripheral blood sample of 100 gastric cancer patients will be collected at the baseline and time point response of therapy.
Procedure: CTC detection — Peripheral blood collected from patients will be administrated to CTC detection.
Procedure: ctDNA detection — DNA extraction from patients' peripheral blood will be measured by 741 panel DNA sequence.
Procedure: 10×genomics single cell RNA sequence — Tissue collected from patients will be digested into single cell suspension and administrated to 10×genomics single cell RNA sequence.
Procedure: Whole exon sequence — DNA will be extracted from patients' tissue and administrated to whole exon sequence.
Procedure: Proteomics detection — Peripheral blood collected from patients will be administrated to proximity extension assay .

SUMMARY:
Dynamic multiomics explore the efficacy and mechanism of anti-HER2 & immunotherapy of HER2 Positive GC

DETAILED DESCRIPTION:
The investigators will recruit 100 HER2 positive advanced gastric cancer patients.Blood and tumor tissue will be collected at treatment baseline, every time point response till disease progression. All samples will be processed by next-generation sequence , 10× genomics single-cell sequence ,whole exon sequence, proteome detection and CTC detection to explore the efficacy and mechanism of anti-HER2 & immunotherapy of HER2 positive GC.

ELIGIBILITY:
Inclusion Criteria:

* Having signed informed consent
* Age:18-80 years old
* HER2 overexpression confirmed by IHC or ISH (IHC 3+,or IHC2+/ISH+)
* Histologically confirmed gastric adenocarcinoma
* Unresectable recurrent or metastatic gastric cancer
* Previous neo-adjuvant or adjuvant treatment for gastric cancer, if applicable, more than 6 months
* Measurable disease according to the RECIST criteria
* Karnofsky performance status ≥70
* Life expectancy of ≥3 month
* No prior radiotherapy except radiotherapy at non-target lesion of the study more than 4 weeks
* ALT and AST<2.5 times ULN (≤5 times ULN in patients with liver metastases)
* Serum albumin level ≥3.0g/dL
* Serum AKP < 2.5 times ULN
* Serum creatinine <ULN, and CCr < 60ml/min
* Bilirubin level < 1.5 ULN
* WBC>3,000/mm3, absolute neutrophil count ≥2000/mm3, platelet>100,000/mm3, Hb>9g/dl

Exclusion Criteria:

* Previous systemic therapy for metastatic gastric cancer
* Surgery (excluding diagnostic biopsy) within 4 weeks prior to study entry Contraindications of nuclear magnetic resonance image such as fitment of cardiac pacemaker , nerve stimulator, or aneurysm clip, and metallic foreign body in eye ball and so on.
* Allergic constitution or allergic history to protium biologic product or any investigating agents.
* Severe heart disease or such history as recorded congestive heart failure, uncontrolled cardiac arrhythmia, angina pectoris needing medication, cardiac valve disease, severe abnormal ECG findings, cardiac infarction , or retractable hypertension.
* Pregnancy or lactation period
* Other previous malignancy within 5 year, except non-melanoma skin cancer
* Legal incapacity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Proportions of HER2 & PD-L1 positive CTC | 2 months
  Numbers of CTC and proportions of HER2 or PD-L1 positive CTC collected at treatment baseline and every time point response will be calculated and recorded. Proportions of HER2 and PD-L1 positive CTC will be compared between two groups.
Incidence rate of ctDNA deletion, amplification, insertion and other types of variation evaluated by next generation sequence(NGS). | 2 months
  NGS will be proceeded to detect the ctDNA variations features at treatment baseline and every time point response will be recorded and compared between two groups.
Proportions of lymphocytes, stromal cells, tumor cells in tumor tissue assessed by single cell transcriptome sequence. | Treatment baseline; Up to 2 months from the initial treatment; From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  single cell digested from tumor tissue will be administrated to 10× genomics single cell transcriptome sequence. Proportions of lymphocytes, stromal cells, tumor cells assessed by single cell transcriptome sequence at treatment baseline, the second time point response and disease progression time point will be recorded and compared between two groups.
Incidence rate of gene deletion, amplification, insertion and other types of variation of tumor evaluated by whole exon sequence(WES). | Treatment baseline; Up to 2 months from the initial treatment; From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  DNA extracted from tumor tissue will be administrated to whole exon sequence.Variation features at treatment baseline, the second time point response and disease progression time point will be recorded and compared between two groups.
Tumor associated proteins expression level of tumor | Treatment baseline; Up to 2 months from the initial treatment; From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  96 tumor associated proteins' expression level of tumor at treatment baseline, second time point response and disease progression time point will be recorded and compared between two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China